CLINICAL TRIAL: NCT04446247
Title: Accuracy of Owlet Smart Sock Sensor 3rd Generation With Profound Hypoxia
Status: Completed | Type: Observational
Sponsor: Owlet Baby Care, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 10-00437
Record Dates: First submitted 2020-06-22; First posted 2020-06-24 (Actual); Results first posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-09

CONDITIONS: Hypoxia
Keywords: Verification of SpO2 accuracy; Induced hypoxia; Owlet Smart Sock; Pulse oximeter
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Owlet Smart Sock Sensor 3rd Generation — Pulse Oximetry

SUMMARY:
Performance testing of pulse oximeters. The protocol involves brief stable arterial oxygen desaturation in healthy volunteers and sampling arterial blood when a stable level of hypoxia has been attained. The blood sample is analyzed for oxygen saturation with a gold standard bench CO-oximeter. This protocol is aligned with the latest ISO and FDA guidance documents for pulse oximeter testing.

ELIGIBILITY:
Inclusion Criteria:

* The subject is male or female, aged ≥18 and <50.
* The subject is in good general health with no evidence of any medical problems.
* The subject is fluent in both written and spoken English.
* The subject has provided informed consent and is willing to comply with the study procedures.

Exclusion Criteria:

* The subject is obese (BMI>30).
* The subject has a known history of heart disease, lung disease, kidney or liver disease.
* Diagnosis of asthma, sleep apnea, or use of CPAP.
* Subject has diabetes.
* Subject has a clotting disorder.
* The subject a hemoglobinopathy or history of anemia, per subject report or the first blood sample, that in the opinion of the investigator, would make them unsuitable for study participation.
* The subject has any other serious systemic illness.
* The subject is a current smoker.
* Any injury, deformity, or abnormality at the sensor sites that in the opinion of the investigators' would interfere with the sensors working correctly.
* The subject has a history of fainting or vasovagal response.
* The subject has a history of sensitivity to local anesthesia.
* The subject has a diagnosis of Raynaud's disease.
* The subject has unacceptable collateral circulation based on exam by the investigator (Allen's test).
* The subject is pregnant, lactating or trying to get pregnant.
* The subject is unable or unwilling to provide informed consent, or is unable or unwilling to comply with study procedures.
* The subject has any other condition, which in the opinion of the investigators' would make them unsuitable for the study.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants in this study should be healthy, between 18 and 50 years of age and willing to participate in breathing studies with or without blood samples in San Francisco.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2020-03-12 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Bickler, MD, Principal Investigator — UCSF Department of Anesthesia; John Feiner, MD, Principal Investigator — UCSF Department of Anesthesia
Locations (1):
- University California San Fransisco, Department of Anesthesia, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- ARMS SpO2 70-100%: Comparison to Reference CO-Oximetry Accuracy of the Owlet Smart Sock Sensor 3rd Generation: The purpose of this study was to validate the SpO2 accuracy of the Owlet Smart Sock Sensor 3rd Generation during non-motion conditions over the range of 70-100% SaO2 as compared to arterial blood samples assessed by CO-Oximetry. It was expected that the Accuracy Root Mean Square (ARMS) performance of the oximetry system would meet the required specification of ARMS of 3.0% or less.
Period: Overall Study
Arm/Group | ARMS SpO2 70-100%
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 14 Healthy volunteer subjects
Units Other Than Participants: Arterial Blood Samples
Arm/Group | ARMS SpO2 70-100%
Number analyzed (Participants) | 14
Number analyzed (Arterial Blood Samples) | 351
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 5
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 14
Skin Tone [Count of Participants; unit: Participants]
  Dark | 1
  Dark-Medium | 4
  Medium | 4
  Light- Medium | 4
  Light | 1

OUTCOME MEASURES:

1. Primary Outcome: SpO2 Accuracy (Arms) of ≤3 Between 70 and 100%
Description: Determination of Average Root Mean Square SpO2 Accuracy of the Owlet Smart Sock 3rd Generation
Time Frame: 1 hour
Measure: Number; unit: Percentage
Units Other Than Participants: Number of Data Points
Groups:
- ARMS SpO2 70-100%, Oximeter #1 (Left): Comparison to Reference CO-Oximetry on the left thumb. Accuracy of the Owlet Smart Sock Sensor 3rd Generation: The purpose of this study was to validate the SpO2 accuracy of the Owlet Smart Sock Sensor 3rd Generation during non-motion conditions over the range of 70-100% SaO2 as compared to arterial blood samples assessed by CO-Oximetry. It was expected that the Accuracy Root Mean Square (ARMS) performance of the oximetry system would meet the required specification of ARMS of 3.0% or less.
- ARMS SpO2 70-100%, Oximeter #2 (Right): Comparison to Reference CO-Oximetry on the right thumb.
  Accuracy of the Owlet Smart Sock Sensor 3rd Generation: The purpose of this study was to validate the SpO2 accuracy of the Owlet Smart Sock Sensor 3rd Generation during non-motion conditions over the range of 70-100% SaO2 as compared to arterial blood samples assessed by CO-Oximetry. It was expected that the Accuracy Root Mean Square (ARMS) performance of the oximetry system would meet the required specification of ARMS of 3.0% or less.
Arm/Group | ARMS SpO2 70-100%, Oximeter #1 (Left) | ARMS SpO2 70-100%, Oximeter #2 (Right)
Number analyzed (Participants) | 14 | 14
Number analyzed (Number of Data Points) | 211 | 247
Percentage | 2.10 | 2.19

ADVERSE EVENTS:
Time Frame: Study Duration (approximately 1 hour)
Description: All subjects completed the study without events.
Groups:
- ARMS SpO2 70-100%, Oximeter #2 (Right): Comparison to Reference CO-Oximetry on the left thumb.
  Accuracy of the Owlet Smart Sock Sensor 3rd Generation: The purpose of this study was to validate the SpO2 accuracy of the Owlet Smart Sock Sensor 3rd Generation during non-motion conditions over the range of 70-100% SaO2 as compared to arterial blood samples assessed by CO-Oximetry. It was expected that the Accuracy Root Mean Square (ARMS) performance of the oximetry system would meet the required specification of ARMS of 3.0% or less.
Arm/Group | ARMS SpO2 70-100%, Oximeter #1 (Left) | ARMS SpO2 70-100%, Oximeter #2 (Right)
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-22): https://cdn.clinicaltrials.gov/large-docs/47/NCT04446247/Prot_SAP_000.pdf